CLINICAL TRIAL: NCT05979220
Title: A Multicenter, Single Arm, Prospective Phase II Clinical Study of Dalpiciclib Combined With Letrozole in the Maintenance Treatment of HR Positive and HER2 Negative Metastatic Breast Cancer After First-line Chemotherapy
Brief Title: Study of Dalpiciclib Combined With Letrozole in the Maintenance Treatment of HR Positive and HER2 Negative Metastatic Breast Cancer After First-line Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shuangyue Liu (Other)
Responsible Party: Sponsor-Investigator, Shuangyue Liu, Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-SC-BC-II-015
Record Dates: First submitted 2023-05-19; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib combined with Letrozole (Experimental): Dalpiciclib combined with Letrozole,28 days as one cycle.
  1. Dalpiciclib: 150 mg (p.o.) was given once daily for 3 weeks, followed by 1 week off in each 4-week cycle.
  2. Letrozole: 2.5mg, p.o., once a day, continuous administration.
  Interventions: Drug: Dalpiciclib combined with Letrozole

INTERVENTIONS:
Drug: Dalpiciclib combined with Letrozole — A multicenter, single arm, prospective Phase II clinical study

SUMMARY:
This study aimed to evaluate the efficacy and safety of Dalpiciclib combined with Letrozole in the maintenance treatment of HR positive and HER2 negative metastatic breast cancer after first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Has the pathologically-confirmed diagnosis of locally recurrent or metastatic, hormone-receptor positive, HER2 negative Breast Cancer.
2. Age: 18 - 75 years old
3. Eastern Cooperative Oncology Group performance status (ECOG PS)=0~1
4. Functions of liver and kidney is normal
5. Agreed to take contraceptive measures during treatment

Exclusion Criteria:

1. Confirmed diagnosis of HER2 positive disease.
2. Central nervous system metastasis
3. Patients who received prior treatment with any CDK4/6 inhibitor.
4. Clinically significant cardiovascular and cerebrovascular diseases,including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention；
5. Researchers believe that is not suitable for the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated up to 23 months
  The time from the enrollment of the subject until the first recording of tumor progression (evaluated according to RECIST 1.1 criteria) or death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival 2(PFS2) | Estimated up to 27-31 months
  The time from the first chemotherapy for the metastatic stage by the subject to the first recording of tumor progression (evaluated according to RECIST 1.1 standards) or death from any cause.

OTHER OUTCOMES:
Overall Survival(OS) | Estimated up to 5 years
  OS was defined as the time from the first study treatment to the date of death from any cause
Objective Response Rate（ORR） | Estimated up to 23 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Clinical Benefit Rate (CBR) | Estimated up to 23 months
  The percentage of participants who received study treatment and evaluated the best overall efficacy according to RECIST 1.1 criteria as complete remission (CR), partial remission (PR), and disease stability (SD) ≥ 24 weeks.
Disease Control Rate (DCR) | Estimated up to 23 months
  Disease Control Rate (DCR) was defined as the percentage of patients with a complete response (CR), partial response (PR) and stable disease (SD).
Patient Reported Outcome (PRO) | Estimated up to 5 years
  Using the European Five Dimensional Health Scale (EQ-5D) to allow patients to self-evaluate their quality of life
Adverse events (AEs) | Estimated up to 5 years
  The drug safety was assessed by investigator(s) according to NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China